CLINICAL TRIAL: NCT02844803
Title: Pilot Study to Investigate the Effect of Metformin and S. Baicalensis Combination Therapy in Type 2 Diabetes Mellitus Patients
Brief Title: Study of Metformin and S. Baicalensis Combination Therapy in Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Namyi Gu (Other)
Responsible Party: Sponsor-Investigator, Namyi Gu, Assistant professor, DongGuk University
Organization: DongGuk University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: S.baicalensis-Metformin
Record Dates: First submitted 2016-07-22; First posted 2016-07-26 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active drug-> Placebo (Other): Metformin + S. Baicalensis --> Metformin + Placebo
  Interventions: Drug: Combination of Metformin + S. Baicalensis; Drug: Combination of Metformin + Placebo
- Placebo -> Active drug (Other): Metformin + Placebo --> Metformin + S. Baicalensis
  Interventions: Drug: Combination of Metformin + S. Baicalensis; Drug: Combination of Metformin + Placebo

INTERVENTIONS:
Drug: Combination of Metformin + S. Baicalensis — the combination therapy for 8 weeks
Drug: Combination of Metformin + Placebo — the metformin single therapy for 8 weeks

SUMMARY:
The study is a pilot trial to investigate the effect of Metformin and S. Baicalensis Combination Therapy in Type 2 Diabetes Mellitus Patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as a diabetes mellitus patient at least 3 months ago on screening
* Treated with metformin of ≥ 500 mg/day over 3 months on screening
* Fasting glucose level of 110~180 mg/dl or HbA1c of 7.0~9.0% on screening

Exclusion Criteria:

* With acute or chronic inflammation
* Treated with systemic corticosteroids within 4 weeks prior to the first administration of study medication
* With heart failure, myocardial infarction, stroke, or other acute severe cardiovascular diseases
* With acute or chronic renal failure or nephrotic syndrome
* With impaired hepatic function.
* Drug or Alcoholic abuser
* Pregnant or nursing woman

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change of serum glucose level after 8 weeks from baseline | Day1 and Day 57 on the 1st and 2nd periods

CONTACTS AND LOCATIONS:
Overall Officials: Han Seok Choi, MD, PhD, Principal Investigator — Dongguk University College of Medicine and Ilsan Hospital
Locations (1):
- Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No